CLINICAL TRIAL: NCT00532194
Title: A Randomised, Placebo-controlled, Trial of Concurrent Cediranib [AZD2171] (With Platinum-based Chemotherapy) and Concurrent and Maintenance Cediranib in Women With Platinum-sensitive Relapsed Ovarian Cancer
Brief Title: An RCT of Concurrent and Maintenance Cediranib in Women With Platinum-sensitive Relapsed Ovarian Cancer
Acronym: ICON6
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Collaborators: Cancer Research UK (Other); National Health and Medical Research Council, Australia (Other); Australia New Zealand Gynaecological Oncology Group (Other); NCIC Clinical Trials Group (Network); Grupo Español de Investigación en Cáncer de Ovario (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Andrew Embleton, ICON6 Statistician, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-001346-41; ISRCTN68510403 (Registry Identifier: ISRCTN); 2007-001346-41 (EudraCT Number); NCT00544973 (obsolete NCT alias)
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; fallopian tube cancer; primary serous peritoneal cancer; gynaecological carcinoma; randomised controlled trial; Cediranib; AZD2171; efficacy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — cediranib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (reference) (Placebo Comparator): Patients in this arm will receive standard platinum based chemotherapy plus a daily oral placebo tablet for the duration of chemotherapy and then until protocol defined disease progression occurs.
- B (concurrent cediranib) (Active Comparator): Patients in this arm will receive standard platinum based chemotherapy plus a daily oral cediranib tablet during chemotherapy only and then an oral daily placebo tablet until protocol defined disease progression occurs.
  Interventions: Drug: cediranib
- C (concurrent and maintenance cediranib) (Active Comparator): Patients in this arm will receive standard platinum based chemotherapy plus a daily oral cediranib tablet during chemotherapy until protocol defined disease progression occurs.
  Interventions: Drug: cediranib

INTERVENTIONS:
Drug: cediranib — Once-daily oral tablet starting dose 20mg
  Other Names: AZD2171; Recentin
  Arms: B (concurrent cediranib); C (concurrent and maintenance cediranib)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of cediranib in combination with standard chemotherapy, in patients who have relapsed with ovarian, fallopian tube or epithelial cancer, after first line platinum based treatment.

DETAILED DESCRIPTION:
ICON6 is a randomised three-arm, two stage, double-blind, placebo-controlled multicentre Gynaecologic Cancer InterGroup (GCIG) phase III trial.

All patients will receive 6 cycles of platinum-based chemotherapy. Trial drug will be administered for up to 18 months from randomisation or until progression, whichever is sooner. Patients who have not progressed at 18 months from randomisation can continue Trial Drug until progression, if in the opinion of the clinician and the patient there is continuing clinical benefit.

Patients in Arm A (the reference arm) will receive a platinum-based chemotherapy regimen plus a daily oral placebo tablet for the duration of the chemotherapy and up to 18 months from randomisation or until progression.

Patients in Arm B (concurrent cediranib arm) will also receive a platinum-based chemotherapy regimen plus daily oral cediranib during chemotherapy only, and then an oral daily placebo tablet up to 18 months from randomisation or until progression.

Patients in Arm C (concurrent and maintenance cediranib arm) will also receive a platinum-based chemotherapy regimen plus oral cediranib daily during chemotherapy and then continued up to 18 months from randomisation or until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged >= 18 years with previous histologically proven diagnosis of

   * Epithelial ovarian carcinoma
   * Fallopian tube carcinoma
   * Primary serous peritoneal carcinoma requiring treatment with further platinum-based chemotherapy > 6 months after their last cycle of first-line chemotherapy and 6 weeks after maintenance that is not chemotherapy based.
2. Signed informed consent and ability to comply with the protocol
3. Ability to commence treatment within approximately 2 weeks of randomisation
4. CT or MRI proven relapsed disease (measurable or non-measurable)
5. ECOG performance status 0-1
6. Life expectancy more than 12 weeks
7. If there is a past history of a solid tumour (other than ovarian cancer), this must have been treated curatively more than five years ago with no evidence of recurrence, with the exception of patients who have synchronous endometrial cancer (stage I G1, G2) with their ovarian cancer
8. If prior anthracycline or chest radiotherapy, Left Ventricular Ejection Fraction (LVEF) > institutional lower limit of normal.
9. Adequate bone marrow function

   * Absolute Neutrophil Count (ANC) >= 1.5 x 109/l
   * Platelets (Plt) >= 100 x 109/l
   * Haemoglobin (Hb) >= 9g/dl (can be post transfusion)
10. Adequate liver function (within 14 days before randomisation)

    * Serum bilirubin (BR) ≤ 1.5 x ULN
    * Serum transaminases ≤ 2.5 x ULN
11. Adequate renal function

    * Serum creatinine ≤ 1.5 ULN or calculated creatinine clearance > 50 ml/min
    * Urine dipstick for proteinuria <2+. If urine dipstick is >= 2+ on two occasions more than one week apart then a 24 hour urine must demonstrate <=1g of protein in 24 hours or protein/creatinine ratio <1.5

Exclusion Criteria:

1. Non-epithelial ovarian cancer, including malignant mixed Mullerian tumours and mucinous carcinoma of the peritoneum
2. Poorly controlled hypertension (persistently elevated > 150/100mmHg, either systolic or diastolic or both, despite anti-hypertensive medication)
3. History of inflammatory bowel disease (Crohn's disease or Ulcerative Colitis)
4. Malignancies other than ovarian cancer within 5 years prior to randomisation, except for synchronous endometrial cancer (Stage I G1,G2) with ovarian cancer,adequately treated carcinoma in situ of the cervix and/or basal cell skin cancer. Patients who have a past history of a solid tumour, treated curatively, more than five years prior to randomisation, with no evidence of recurrence, are still eligible to enter ICON6.
5. Previous radiotherapy within 21 days prior to anticipated start of treatment
6. Treatment with any other investigational agent within 6 weeks prior to entering this trial. Patients are still eligible for entry into ICON6 if they have received previous treatment for ovarian cancer with either bevacizumab, erlotinib, or a Cox-2 inhibitor as long as more than 6 weeks have elapsed since the last treatment.
7. Arterial thrombotic event (including transient ischaemic attack [TIA], cerebrovascular accident [CVA) and peripheral arterial embolus) within the previous 12 months.
8. GI impairment that could affect ability to take, or adsorption of, oral medicines including sub acute or complete bowel obstruction
9. Known hypersensitivity to cediranib or other VEGF inhibitors
10. Major surgery within 2 weeks before anticipated start of treatment
11. Significant haemorrhage of > 30ml in a single episode within 3 months or any haemoptysis
12. Evidence of severe or uncontrolled cardiac disease

    * Myocardial infarct [MI] or unstable angina within 12 months
    * New York Health Association (NYHA) ≥ grade 2 congestive heart failure (CHF)
    * Cardiac ventricular arrhythmias requiring medication.
    * History of 2nd or 3rd degree atrioventricular conduction defects.
13. Prolonged QTc (corrected) interval of > 470msec on ECG, or a family history of long QT syndrome.
14. Persisting ≥ Grade 2 CTC toxicity (except alopecia and neuropathy) from previous anti-cancer treatment. If peripheral sensory or motor neuropathy ≥ grade 2 then paclitaxel can be omitted from the chemotherapy at the discretion of the treating physician
15. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory in the case of suspected brain metastases. Spinal MRI is mandatory in the case of suspected spinal cord compression. Patients with unstable, untreated brain or meningeal metastases are not eligible.
16. Inability to attend or comply with treatment or follow-up scheduling
17. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
18. Fertile women of childbearing potential not willing to use adequate contraception for the duration of trial treatment and at least 6 months after.
19. Any other severe uncontrolled medical condition or disease
20. Concomitant use of potent inhibitors of CYP3A4 and 2C8 which cannot be stopped without a 2 week washout period before starting Trial Drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2007-07; Primary Completion 2013-04 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Apr 2013

SECONDARY OUTCOMES:
Overall survival | Q2 2016
Toxicity | Q2 2015
Quality of Life | Q2 2015

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ledermann, Prof., Principal Investigator — University College, London
Locations (1):
- University College London, London, Greater London, United Kingdom

REFERENCES:
- [Background] Raja FA, Griffin CL, Qian W, Hirte H, Parmar MK, Swart AM, Ledermann JA. Initial toxicity assessment of ICON6: a randomised trial of cediranib plus chemotherapy in platinum-sensitive relapsed ovarian cancer. Br J Cancer. 2011 Sep 27;105(7):884-9. doi: 10.1038/bjc.2011.334. Epub 2011 Aug 30. PMID 21878941
- [Result] Ledermann J, Perren T, Raja F, Embleton A, Rustin GJS, Jayson G, Kaye SB, Swart AM, Vaughan M, Hirte H. Randomised double-blind phase III trial of cediranib (AZD 2171) in relapsed platinum sensitive ovarian cancer: Results of the ICON6 trial. Eur J Cancer 2013;49(Suppl. 3):S5 (LBA10).
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Ledermann JA, Embleton-Thirsk AC, Perren TJ, Jayson GC, Rustin GJS, Kaye SB, Hirte H, Oza A, Vaughan M, Friedlander M, Gonzalez-Martin A, Deane E, Popoola B, Farrelly L, Swart AM, Kaplan RS, Parmar MKB; ICON6 collaborators. Cediranib in addition to chemotherapy for women with relapsed platinum-sensitive ovarian cancer (ICON6): overall survival results of a phase III randomised trial. ESMO Open. 2021 Apr;6(2):100043. doi: 10.1016/j.esmoop.2020.100043. Epub 2021 Feb 18. PMID 33610123
- [Derived] Ledermann JA, Embleton AC, Raja F, Perren TJ, Jayson GC, Rustin GJS, Kaye SB, Hirte H, Eisenhauer E, Vaughan M, Friedlander M, Gonzalez-Martin A, Stark D, Clark E, Farrelly L, Swart AM, Cook A, Kaplan RS, Parmar MKB; ICON6 collaborators. Cediranib in patients with relapsed platinum-sensitive ovarian cancer (ICON6): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2016 Mar 12;387(10023):1066-1074. doi: 10.1016/S0140-6736(15)01167-8. PMID 27025186